CLINICAL TRIAL: NCT07288307
Title: Ultrasound Guided Surgical Evacuation Versus Combined Local and Systemic Methotrexate Injection for Management of Caesarean Scar Pregnancy [Clinical Trial ]
Brief Title: Surgical Evacuation Versus Methotrexate Injection in Treatment of Caesarean Scar Pregnancy [Clinical Trial ]
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Badr Atef Abd Allah Moussa, Badr Atef, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-MTX-01
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Caesarean Scar Pregnancy
MeSH Terms: interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound surgical evacuation (Experimental)
  Interventions: Procedure: Surgical evacuation and methotrexate injection
- Local and systemic methotrexate injection (Active Comparator)
  Interventions: Procedure: Surgical evacuation and methotrexate injection

INTERVENTIONS:
Procedure: Surgical evacuation and methotrexate injection — Surgical evacuation of the scar pregnancy using ultrasound and local and systemic methotrexate injection

SUMMARY:
The aim of the study is to compare the effectiveness and the complications of Ultrasound guided surgical evacuation versus using combined local and systemic methotrexate injection for management of caesarean scar pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Gestation age Less than 12 weeks. Hemodynamically stable patient with un ruptured CSP. Non disturbed scar pregnancy . Acceptance of possible prolonged follow up, repeated HCG tests, the need for additional treatment doses and possible bleeding and subsequent hysterectomy.

-

Exclusion Criteria:

* Patient refuse TOP. Gestation age More than 12 weeks . Hemodynamically unstable patient with ruptured CSP. Contraindication for methotrexate as hepatic disorders, renal disorders ,hypersensitivity to the drug and autoimmune diseases.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of treatment either by surgical evacuation or by methotrexate injection | Up to 8 weeks post -intervention
  The proportion of participants achieving complete resolution of caesarean scar pregnancy without the need of additional intervention

SECONDARY OUTCOMES:
Bleeding during the procedure | Up to 8 weeks post -intervention
The need for additional intervention | Up to 8 weeks post -intervention
Time for serum-hCG normalisation (days). | Up to 8 weeks post -intervention
Hospital stay (days). | Up to 8 weeks post -intervention
Uterine perforation. | Up to 8 weeks post -intervention
Occurrence of drug complications | Up to 8 weeks post -intervention

REFERENCES:
- [Background] Larsen JV, Solomon MH. Pregnancy in a uterine scar sacculus--an unusual cause of postabortal haemorrhage. A case report. S Afr Med J. 1978 Jan 28;53(4):142-3. PMID 653492
- [Background] Seow KM, Huang LW, Lin YH, Lin MY, Tsai YL, Hwang JL. Cesarean scar pregnancy: issues in management. Ultrasound Obstet Gynecol. 2004 Mar;23(3):247-53. doi: 10.1002/uog.974. PMID 15027012
- [Background] Jurkovic D, Hillaby K, Woelfer B, Lawrence A, Salim R, Elson CJ. First-trimester diagnosis and management of pregnancies implanted into the lower uterine segment Cesarean section scar. Ultrasound Obstet Gynecol. 2003 Mar;21(3):220-7. doi: 10.1002/uog.56. PMID 12666214
- [Background] Rotas MA, Haberman S, Levgur M. Cesarean scar ectopic pregnancies: etiology, diagnosis, and management. Obstet Gynecol. 2006 Jun;107(6):1373-81. doi: 10.1097/01.AOG.0000218690.24494.ce. PMID 16738166
- [Background] Qian ZD, Guo QY, Huang LL. Identifying risk factors for recurrent cesarean scar pregnancy: a case-control study. Fertil Steril. 2014 Jul;102(1):129-134.e1. doi: 10.1016/j.fertnstert.2014.04.003. Epub 2014 May 10. PMID 24825421
- [Background] Maymon R, Halperin R, Mendlovic S, Schneider D, Herman A. Ectopic pregnancies in a Caesarean scar: review of the medical approach to an iatrogenic complication. Hum Reprod Update. 2004 Nov-Dec;10(6):515-23. doi: 10.1093/humupd/dmh042. Epub 2004 Sep 16. PMID 15375087
- [Background] Yang MJ, Jeng MH. Combination of transarterial embolization of uterine arteries and conservative surgical treatment for pregnancy in a cesarean section scar. A report of 3 cases. J Reprod Med. 2003 Mar;48(3):213-6. PMID 12698784
- [Background] Peng KW, Lei Z, Xiao TH, Jia FG, Zhong WX, Gao Y, Shen BX, Xie JW. First trimester caesarean scar ectopic pregnancy evaluation using MRI. Clin Radiol. 2014 Feb;69(2):123-9. doi: 10.1016/j.crad.2013.07.021. Epub 2013 Dec 6. PMID 24315547
- [Background] Vial Y, Petignat P, Hohlfeld P. Pregnancy in a cesarean scar. Ultrasound Obstet Gynecol. 2000 Nov;16(6):592-3. doi: 10.1046/j.1469-0705.2000.00300-2.x. No abstract available. PMID 11169360
- [Background] Weimin W, Wenqing L. Effect of early pregnancy on a previous lower segment cesarean section scar. Int J Gynaecol Obstet. 2002 Jun;77(3):201-7. doi: 10.1016/s0020-7292(02)00018-8. PMID 12065130